CLINICAL TRIAL: NCT06581081
Title: Bridging Allogeneic Hematopoietic Stem Cell Transplantation or Not After CD19 CAR - T (S1904) Cell Therapy for r/r B-cell Acute Lymphoblastic Leukemia, a Prospective, Open, Multicenter, Randomized, Control Study (COMPLETE Study)
Brief Title: Bridging Allogeneic Hematopoietic Stem Cell Transplantation or Not After CD19 CAR - T (S1904) Cell Therapy for r/r B-cell Acute Lymphoblastic Leukemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: The First Affiliated Hospital of Soochow University (Other); Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Xiao-Jun Huang, Prof., Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMPLETE
Record Dates: First submitted 2024-08-29; First posted 2024-08-30 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Relapsed Adult ALL; B-cell Acute Lymphoblastic Leukemia; Refractory Acute Lymphoblastic Leukemia; Relapsed Pediatric ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bridging to allo-HSCT (Experimental): Subjects enrolled in this study will first receive Senl_B19 autologous CAR-T (S1904) treatment. If the subject achieves bone marrow leukemia-free state (MLFS) and minimal residual disease (MRD) negative within 12 weeks after S1904 infusion, they will be randomly assigned to the bridging transplant group and the non-bridging transplant group at a ratio of 2:1.
  Interventions: Biological: Senl_B19 autologous CAR-T (S1904) treatment
- No bridging to allo-HSCT (Other): Subjects enrolled in this study will first receive Senl_B19 autologous CAR-T (S1904) treatment. If the subject achieves bone marrow leukemia-free state (MLFS) and minimal residual disease (MRD) negative within 12 weeks after S1904 infusion, they will be randomly assigned to the bridging transplant group and the non-bridging transplant group at a ratio of 2:1.
  Interventions: Biological: Senl_B19 autologous CAR-T (S1904) treatment

INTERVENTIONS:
Biological: Senl_B19 autologous CAR-T (S1904) treatment — Subjects enrolled in this study will first receive Senl_B19 autologous CAR-T (S1904) treatment.

SUMMARY:
Traditional salvage chemotherapy has low efficacy and poor long-term prognosis for relapsed or refractory (R/R) B-cell acute lymphoblastic leukemia (B-ALL). Targeted CD19 CAR-T cell immunotherapy is an effective means of treating R/R B-ALL. Several clinical studies have shown that its remission rate for R/R B-ALL can reach 68-93%. However, long-term follow-up found that the remission time after CD19 CAR-T treatment is short and the relapse rate is high. Therefore, how to ensure the long-term survival of R/R B-ALL patients after remission by CAR-T therapy is an urgent problem to be solved. Some studies have shown that timely bridging allo-HSCT after CAR-T treatment can overcome the risk of relapse and further improve the long-term survival of patients. However, there is currently no randomized controlled study on whether to bridge transplantation after CAR-T. The purpose of this study is to evaluate the efficacy and safety of S1904 in the treatment of relapsed or refractory CD19-positive B-cell acute lymphoblastic leukemia with or without bridging to allogeneic hematopoietic stem cell transplantation after remission.

ELIGIBILITY:
Inclusion Criteria:

1. The subject or guardian understands and voluntarily signs the Informed Consent Form (ICF);
2. Male or female, aged 12-65 years (including the cutoff value) when signing the informed consent form;
3. Expected survival period is not less than 12 weeks;
4. ECOG physical performance score is 0-1 when signing the ICF;
5. The subject must be diagnosed with relapsed/refractory B-cell acute lymphoblastic leukemia when signing the ICF, and at least one of the following must be met:

   1. Relapse: including relapse within 12 months after the first remission, 2 or more relapses;
   2. Refractory: including primary refractory, failure to achieve remission after at least 2 courses of induction therapy, or failure to achieve remission after at least 1 course of salvage therapy after the first relapse.
6. For patients with Philadelphia chromosome-positive ALL (Ph+ ALL), in addition to meeting the above relapse or refractory criteria, they should have failed at least two tyrosine kinase inhibitor (TKI) treatments (except for those with T315I mutations), or be unable to tolerate TKI treatment, or have contraindications to TKI treatment;
7. Bone marrow morphology examination at screening showed that the proportion of primitive immature lymphocytes in the bone marrow was >5%;
8. Tumor cells in the bone marrow or peripheral blood were CD19 positive by flow cytometry at screening;
9. Major organ functions must meet the following requirements:

   1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×upper limit of normal (ULN);
   2. Total bilirubin ≤2×ULN;
   3. Serum creatinine clearance of adult subjects ≥60 mL/min (Cockcroft-Gault formula) or creatinine ≤1.5×upper limit of normal (ULN);
   4. Serum creatinine for children: no more than 1.2 mg/dL for 10 to 13 years old, no more than 1.5 mg/dL for males aged 13 to 16 years old, no more than 1.4 mg/dL for females aged 13 years and above, and no more than 1.7 mg/dL for males aged 16 years and above.
10. Blood oxygen saturation>92%;
11. Males and females of childbearing age with fertility must agree to use effective contraceptive measures from the signing of the informed consent form until 2 years after the use of the study drug. Females of childbearing age include premenopausal women and women within 2 years after menopause. The blood pregnancy test of females of childbearing age must be negative at the time of screening.

Exclusion Criteria:

1. Isolated extramedullary relapse;
2. Burkitt's lymphoma/leukemia;
3. Previous history of CNS disease, including but not limited to epilepsy, paralysis, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, neuropathy (except inactive CNS leukemia);
4. Previous hematopoietic stem cell transplantation;
5. History of autoimmune disease requiring systemic immunosuppressive drug treatment within 2 years before signing the ICF (including but not limited to Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus, systemic sclerosis, inflammatory bowel disease, vasculitis, psoriasis);
6. Any uncontrolled active infection at the time of signing the ICF or within 4 weeks before apheresis, requiring antibiotic, antiviral or antifungal treatment;
7. Previous cell therapy targeting CD19 (autologous or allogeneic);
8. Received CAR-T therapy or other cell/gene therapy before screening;
9. Those who tested positive for hepatitis B surface antigen (HBsAg) during screening need to be excluded; if HBsAg is negative but hepatitis B core antibody (HBcAb) is positive, those with peripheral blood hepatitis B virus (HBV) DNA above the detection limit need to be excluded; those who tested positive for hepatitis C virus (HCV) antibody and HCV RNA need to be excluded; those who tested positive for human immunodeficiency virus (HIV) antibody; those who tested positive for cytomegalovirus (CMV) DNA; those who tested positive for human lymphotropic herpes virus (EBV) DNA; those who tested positive for both Treponema pallidum-specific and non-specific antibodies;
10. Clinically significant cardiovascular disease, including any of the following:

    1. QTc interval ≥470 ms after heart rate correction (QTc interval calculated by Fridericia formula);
    2. New York Heart Association (NYHA) grade II or above heart failure;
    3. Unstable angina or acute myocardial infarction within 6 months before signing the ICF;
    4. Left ventricular ejection fraction (LVEF) < 50%;
    5. Poorly controlled hypertension (systolic blood pressure ≥ 150 mm Hg and/or diastolic blood pressure ≥ 95 mm Hg);
    6. Arrhythmias with clinical significance or requiring antiarrhythmic treatment (such as sustained ventricular tachycardia, ventricular fibrillation, torsade de pointes tachycardia and complete left bundle branch block, etc.);
11. Allergic to any drug component to be used in this study, including but not limited to S1904, clearing drugs (cyclophosphamide, fludarabine), etc.;
12. Received any study drug treatment or other systemic anti-tumor treatment within 4 weeks before apheresis (or 5 half-lives of the drug, whichever is more appropriate as determined by the researcher);
13. Received extensive radiotherapy within 4 weeks before signing the ICF, except for local radiotherapy of non-target lesions for symptom relief within 2 weeks before signing the ICF or expected during the study period;
14. At the time of signing the ICF, except for alopecia and pigmentation, the toxicity caused by previous anti-tumor treatment has not recovered to grade 1 or baseline level (according to NCI-CTCAE version 5.0);
15. Patients who need to receive systemic corticosteroids (dose equivalent to or higher than 10 mg/day of prednisone) or other immunosuppressive drugs within 2 weeks before signing the ICF or within 2 weeks before apheresis or during the study, except for the following:

    1. Intranasal, inhaled, local steroids or local steroid injections (such as intra-articular injections), or
    2. Systemic corticosteroid treatment not exceeding 10 mg/day of prednisone or its equivalent physiological dose, or
    3. Steroids as a preventive medication for allergic reactions (such as pretreatment before computed tomography [CT]), or
    4. Used for symptomatic treatment of adverse reactions after reinfusion;
16. Subjects who have undergone major surgery (except routine biopsy) within 4 weeks before signing the ICF, or are expected to undergo major surgery during the study;
17. Subjects with a history of active tuberculosis infection within 1 year before signing the ICF (except for subjects with a history of active tuberculosis infection more than 1 year ago who are judged by the investigator to have no evidence of active tuberculosis);
18. Subjects with clinically significant thyroid dysfunction as judged by the investigator;
19. Subjects with or with a history of interstitial lung disease or interstitial pneumonia;
20. Subjects with a history of other primary malignant tumors within 5 years before signing the ICF, except for the following:

    1. Cervical carcinoma in situ that has been fully treated and cured;
    2. Localized basal cell carcinoma or squamous cell carcinoma of the skin;
21. Subjects who have received attenuated/inactivated vaccines within 4 weeks before signing the ICF, or subjects who are planned to receive attenuated/inactivated vaccines during the screening period;
22. The researcher believes that the subject's complications or other conditions may affect compliance with the protocol or may be unsuitable for participation in this study;
23. Pregnancy or lactation.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
2-year event-free survival after randomization | Participants will be followed for an expected average of 2 years
  The time from randomization to MRD positive or relapse or death due to non-relapse causes (whichever occurs first)

SECONDARY OUTCOMES:
2-year relapse-free survival after randomization | Participants will be followed for an expected average of 2 years
  Time from randomization to relapse or death from any cause (whichever occurs first)
Cumulative incidence of relapse | Participants will be followed for an expected average of 2 years
  Time from randomization to relapse
2-year overall survival after randomization | Participants will be followed for an expected average of 2 years
  Time from randomization to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People'S Hospital, Beijing, Beijing Municipality, China